CLINICAL TRIAL: NCT07222345
Title: Feasibility of High Intensity Interval Training in Survivors of Childhood, Adolescent, and Young Adult Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FITHOD
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin Lymphoma
Keywords: Childhood Cancer Survivor
MeSH Terms: conditions — Hodgkin Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT Intervention Group (Experimental): Participants will complete a 12-week HIIT program with three 25-minute sessions per week. Each session includes warm-up, five cycles of high-intensity intervals (80-95% peak HR) and recovery periods (50-60% peak HR), and cool-down.
  Interventions: Behavioral: High Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — Participants will complete a 12-week HIIT program with three 25-minute sessions per week. Each session includes warm-up, five cycles of high-intensity intervals (80-95% peak HR) and recovery periods (50-60% peak HR), and cool-down.

SUMMARY:
This pilot study evaluates the feasibility of a 12-week high intensity interval training (HIIT) program in survivors of childhood, adolescent, and young adult Hodgkin lymphoma within 24 months of completing treatment. Preliminary efficacy of the HIIT intervention for improved cardiorespiratory fitness, body composition, physical function, autonomic response to exercise, peripheral neuropathy, biological aging markers, and physical activity will also be evaluated.

Primary Objective:

To determine the feasibility of a 12-week high intensity interval training (HIIT) program in survivors of childhood, adolescent, and young adult Hodgkin lymphoma within 24 months of completing treatment.

Feasibility will be assessed by:

* Participation Rate: Number of eligible survivors approached who enroll.
* Completion Rate: Number of scheduled HIIT sessions attended and number of enrolled participants who complete post-intervention testing.

DETAILED DESCRIPTION:
Hodgkin lymphoma survivors face elevated risks of cardiovascular disease and premature aging. HIIT, which alternates high-intensity effort with recovery periods, has shown benefits in adult cancer survivors but has not been tested in younger populations. This study will assess whether recently treated survivors can complete a remotely supervised 12-week HIIT program and evaluate its effects on multiple health outcomes. Participants will undergo baseline and post-intervention assessments including exercise testing, body composition, autonomic function, and blood biomarkers. The intervention is delivered via a secure web-based platform with live supervision by exercise physiologists.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with Hodgkin lymphoma between the ages of 10 to 25 years.
* Participant is between the ages of >10 and <25 years old the time of enrollment.
* Participant has completed treatment (end of chemotherapy for those not receiving radiation therapy or end of radiation therapy) for Hodgkin lymphoma within 24 months prior to enrollment and recovered from any acute treatment-related adverse events.
* Participant has been medically cleared to participate in physical activity.
* Participant verbalizes understanding of directions for use of the web-based platform on the study provided iPad and heart rate monitor.

Exclusion Criteria:

* Participant has evidence of relapsed disease.
* Participant has a diagnosis of acute heart failure.
* Participant reports currently participating in HIIT training or >420 minutes per week of moderate to vigorous physical activity.
* Female participant who is currently pregnant.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate (percent of eligible participants approached who enroll) | Trial completion (12 weeks)
  Descriptive statistics will be reported
Completion rate (percentage of scheduled HIIT sessions attended and percentage of post-intervention testing sessions completed) | Trial completion (12 weeks)
  Descriptive statistics will be reported

OTHER OUTCOMES:
Cardiorespiratory fitness (VO2peak, ml/kg/min) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Ewing battery score of autonomic function (0 to 5 points) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Body mass index (weight and height will be combined to report body mass index in kg/m2) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Percent body fat (%) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Lean mass percentage (%) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Visceral fat level (score) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Hand grip strength (kg) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Knee extension strength (N/kg) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Modified total neuropathy scale (0 to 24 points) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
DNA methylation | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Mitochondrial DNA copy number | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Telomere length (kb) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
High-sensitivity C-reactive protein (mg/L) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Interleukin-6 (pg/mL) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported
Physical activity (kilocalories per week) | baseline at study entry, 12 weeks
  Descriptive statistics of the change between baseline and 12 weeks will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Amy Berkman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols